CLINICAL TRIAL: NCT02126540
Title: A Non-randomized, Multi-center Feasibility Trial of the Avinger Pantheris System, an Atherectomy Device That Provides Directional Visualization and Imaging While Removing Plaque in Diseased Lower Extremity Arteries
Brief Title: Trial of Pantheris System, an Atherectomy Device That Provides Imaging While Removing Plaque in Lower Extremity Arteries
Acronym: COMBINE-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0638
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease; Atherectomy; Optical Coherence Tomography
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary Cohort (Experimental): Main cohort; treatment Arm with Pantheris Atherectomy System
  Interventions: Device: Pantheris Atherectomy System

INTERVENTIONS:
Device: Pantheris Atherectomy System — Treatment device in primary cohort arm; OCT image guided directional atherectomy
  Other Names: Pantheris

SUMMARY:
To evaluate the safety and effectiveness of the Pantheris System to perform atherectomy while using directional visualization and imaging as an adjunct to fluoroscopy to aid removal of plaque from diseased lower extremity arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patient is a candidate for percutaneous intervention for peripheral vascular disease in the legs.
3. Patient is willing and able to give informed consent
4. Documented symptomatic atherosclerotic peripheral vascular disease Rutherford Classification 2-5.
5. Reference vessel lumen proximal to target lesion >3.0 mm in diameter by visual estimation.
6. Subject has de novo target lesion(s) with stenosis >70% by visual estimation distal to the profunda femoral artery. No more than 2 lesions may be treated with the Pantheris device.
7. Target lesion length <10 cm if target lesion >70% and <99% stenosed. If target lesion a chronic total occlusion (99-100% stenosed), target lesion length <4 cm.
8. Patient is capable of meeting requirements and be present at the follow-up clinic visits at 30 days.
9. At least one patent tibial run-off vessel at baseline. -

Exclusion Criteria:

1. Subject is pregnant or breast feeding.
2. Rutherford Class 0 to 1 (asymptomatic and mild claudication).
3. Rutherford Class 6 (critical limb ischemia).
4. Severe calcification of the target lesion.
5. Target lesion with any type of stent or graft.
6. Target lesion in the iliac artery.
7. Target lesion stenosis <70%.
8. Subjects with significant (>70%) occlusive lesions proximal to the target lesion not successfully treated during the index procedure (upstream disease) and prior to treatment of the target lesion.
9. Endovascular or surgical procedure performed on the index limb less than or equal to 30 days prior to the index procedure.
10. Planned endovascular or surgical procedure 30 days after the index procedure.
11. Lesion in the contralateral limb requiring intervention during the index procedure or within 30 days of the index procedure.
12. Subjects with active infections whether they are being currently treated or not.
13. Hemodialysis or GFR <30 mL/min or creatinine level >2.5mg/dL.
14. Evidence or history of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months.
15. Evidence or history of aneurysmal target vessel within the past 2 months.
16. History of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
17. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
18. Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated.
19. History of heparin-induced thrombocytopenia (HIT).
20. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/mm2 , known coagulopathy, or INR >1.5.
21. Any thrombolytic therapy within 2 weeks of the index procedure.
22. Any clinical and/or angiographic complication attributed to the use of another device prior to the insertion of the Pantheris into the subject.
23. Subjects or their legal guardians who have not or will not sign the Informed Consent.
24. Subjects who are unwilling or unable to comply with the follow-up study requirements.
25. Participation in any study of an investigational device, medication, biologic or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint | Day 0 through Day 30
  The primary safety endpoint is defined as freedom from major adverse events (MAE) through 30 day follow-up:
  * Clinically driven target lesion revascularization (TLR)
  * Myocardial infarction (MI)
  * Cardiovascular related deaths
  * Unplanned, major index limb amputation
  * Device Related Events:
    * Clinically Significant Perforations
    * Clinically Significant Dissections
    * Clinically Significant Embolus
    * Pseudoaneurysm
Primary Effectiveness Endpoint | Day 0
  The primary efficacy endpoint of technical success is defined as the percent of target lesions that has a residual diameter stenosis <50% post the Pantheris device alone as assessed by an independent review at the time of treatment using quantitative angiography or visual estimate.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | Day 0
  Freedom from procedural emboli, defined as a new occlusion of any visualized runoff vessel which cannot be reversed with an intravascular vasodilator.
Secondary Effectiveness Endpoint | Day 0
  Procedural success defined as the percent of target lesions that have residual diameter stenosis < 30% post-Pantheris and any other adjunctive therapy.
Secondary Effectiveness Endpoint | Day 30
  Ankle-Brachial Index at 30 days
Secondary Effectiveness Endpoint | Day 30
  Rutherford Classification at 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Andreq Holden, MD, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand